CLINICAL TRIAL: NCT04963010
Title: Impact of Second Forward View Examination of the Proximal Colon on Adenoma Detection Rate
Brief Title: Impact of SFV of Proximal Colon on ADR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Xiaojia (Other)
Responsible Party: Sponsor-Investigator, Zhu Xiaojia, Attending physician, Third People's Hospital of Jingdezhen City
Organization: Third People's Hospital of Jingdezhen City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ThirdPeoplesHJingdezhenCity
Record Dates: First submitted 2021-06-15; First posted 2021-07-15 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Adenoma Detection Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard withdrawal colonoscopy (No Intervention): Observation of conventional colonoscopy
- second forward view (Experimental): second forward view examination of the proximal colon
  Interventions: Diagnostic Test: second forward view

INTERVENTIONS:
Diagnostic Test: second forward view — second forward view examination of the proximal colon
  Arms: second forward view

SUMMARY:
To evaluate the impact of second forward view examination of the proximal colon on adenoma detection rate Inclusion criteria：Patients ≥18 years of age undergoing screening, follow-up monitoring, and diagnostic colonoscopy Exclusion criteria：①Cecal intubation failed. ②Have a history of colorectal surgery. ③Insufficient bowel preparation, inadequate bowel preparation quality (Boston Bowel Preparation Scale (BBPS)scores < 2 in any segment of the colon). ④Inflammatory bowel disease or intestinal tuberculosis. ⑤Familial polyp syndrome. ⑥polyp retrieval failure. ⑦Patients with coagulation dysfunction.

Patients ≥ 18 years of age who came to our hospital's Digestive Endoscopy Center for screening, follow-up monitoring and diagnosis of colonoscopy. After successfully insert the cecum, colonoscope withdrawal to the splenic flexure, all polyps found during the withdrawal process were resection,then they were randomized to standard withdrawal colonoscopy or second forward view according to the random number table (1:1) to perform.

DETAILED DESCRIPTION:
Background:

Colonoscopy can reduce the incidence and mortality rates of colorectal cancer, and the reduction in distal colon cancer is more pronounced than proximal colon cancer. Compared with CRC found on screening, interphase CRC is more likely to occur in the proximal colon above the splenic flexure. Adenoma detection rate (ADR) is an important quality indicator of colonoscopy. Compared with ADR>20%，the incidence of interphase CRC is 10 times higher for endoscopists with ADR<20%. For every 1% increase in ADR, the risk of interphase CRC can be reduced by 3%, and fatal interphase CRC can be reduced by 5%. It is reported in the literature that the second forward view examination of the right colon (cecum, ascending colon, liver flexure) can significantly improve the right colon ADR, however, there is no report on the impact of second forward view examination of the proximal colon ADR (cecum, ascending colon, liver flexure, and transverse colon).

Objective:

To evaluate the impact of second forward view examination of the proximal colon on adenoma detection rate Inclusion criteria： Patients ≥18 years of age undergoing screening, follow-up monitoring, and diagnostic colonoscopy Exclusion criteria：

①Cecal intubation failed. ②Have a history of colorectal surgery. ③Insufficient bowel preparation, inadequate bowel preparation quality (Boston Bowel Preparation Scale (BBPS)scores < 2 in any segment of the colon). ④Inflammatory bowel disease or intestinal tuberculosis. ⑤Familial polyp syndrome. ⑥polyp retrieval failure. ⑦Patients with coagulation dysfunction.

Methods:

Patients ≥ 18 years of age who came to our hospital's Digestive Endoscopy Center for screening, follow-up monitoring and diagnosis of colonoscopy. After successfully insert the cecum, colonoscope withdrawal to the splenic flexure, all polyps found during the withdrawal process were resection,then they were randomized to standard withdrawal colonoscopy or second forward view according to the random number table (1:1) to perform.

Primary Outcome:

proximal colon adenoma detection rate：proportion of patients with proximal colon adenoma found in all colonoscopy patients Secondary Outcome whole colon adenoma detection rate：proportion of patients with colonic adenoma found in all colonoscopy patients Cecal insertion time: the time elapsed from introducing the colonoscope into the anus until intubation of the cecum.

proximal colon withdrawal time: observation time of proximal colon in the absence of polyp removal total withdrawal time:the time measured from when the colonoscope reaches the cecum to the time the scope is withdrawn from the anus in the absence of polyp removal BBPS：Boston bowel preparation score whole colon polyp detection rate：proportion of patients with colonic polyp found in all colonoscopy patients proximal colon polyp detection rate：proportion of patients with proximal colon polyp found in all colonoscopy

Research design Patients ≥ 18 years of age who came to our hospital's Digestive Endoscopy Center for screening, follow-up monitoring and diagnosis of colonoscopy. After successfully insert the cecum, colonoscope withdrawal to the splenic flexure, all polyps found during the withdrawal process were resection,then they were randomized to standard withdrawal colonoscopy or second forward view according to the random number table (1:1) to perform. Patients in the second forward view (SFV) group were inserted into the cecum again , colonoscope withdrawal to the splenic flexure, and the newly discovered polyps in the second forward view were also resection. Patients in the standard withdrawal colonoscopy withdraw the scope from the splenic flexure until exiting the anus,observe, if polyps are found, undergo endoscopic resection.

The assistant is responsible for recording the time.Cecal insertion time refers to the time elapsed from introducing the colonoscope into the anus until intubation of the cecum. Proximal colon withdrawal time refers to the observation time of proximal colon. And the total withdrawal time refers to the time measured from when the colonoscope reaches the cecum to the time the scope is withdrawn from the anus in the absence of polyp removal. Record BBPS, the number, location, size, Paris type and postoperative pathology of polyps.

ELIGIBILITY:
Inclusion Criteria:Patients ≥18 years of age undergoing screening, follow-up monitoring, and diagnostic colonoscopy -

Exclusion Criteria:①Cecal intubation failed. ②Have a history of colorectal surgery. ③Insufficient bowel preparation, Boston Bowel Preparation Score (BBPS) <6 points. ④Inflammatory bowel disease or intestinal tuberculosis. ⑤Familial polyp syndrome. ⑥Recovery of polyp specimens failed, and no histopathological data. ⑦Patients with coagulation dysfunction.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-06-08 (Estimated); Study Completion 2022-06-08 (Estimated)

PRIMARY OUTCOMES:
proximal colon adenoma detection rate | up to 2 years
  proportion of patients with proximal colon adenoma found in all colonoscopy patients

SECONDARY OUTCOMES:
whole colon adenoma detection rate | up to 2 years
  proportion of patients with colonic adenoma found in all colonoscopy patients
Cecal insertion time | up to 2 years
  the time elapsed from introducing the colonoscope into the anus until intubation of the cecum
proximal colon withdrawal time | up to 2 years
  observation time of proximal colon in the absence of polyp removal
total withdrawal time | up to 2 years
  the time measured from when the colonoscope reaches the cecum to the time the scope is withdrawn from the anus in the absence of polyp removal
BBPS | up to 2 years
  Boston bowel preparation score
whole colon polyp detection rate | up to 2 years
  proportion of patients with colonic polyp found in all colonoscopy patients
proximal colon polyp detection rate | up to 2 years
  proportion of patients with proximal colon polyp found in all colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, Study Director — Third People's Hospital of Jingdezhen City
Locations (1):
- Third People's Hospital of Jingdezhen City, Jingdezhen, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Sharing data after the research over
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Half a year after the research over and lasts for 2 years
Access Criteria: Gastroenterologist
URL: http://www.clinicaltrials.gov